CLINICAL TRIAL: NCT00404690
Title: Bedside Silo Versus Attempted Operative Closure for Gastroschisis: A Pilot Study
Brief Title: Bedside Silo Versus Operative Closure for Gastroschisis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in referral pattern changed the population we were studying
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06 09 141
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Gastroschisis
Keywords: Gastroschisis; Silo; Operative closure
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Operative attempt at closure
  Interventions: Procedure: Operative attempt at closure
- 2 (Experimental): bedside silo
  Interventions: Procedure: Bedside Silo

INTERVENTIONS:
Procedure: Bedside Silo — silo placed at bedside on admission
  Arms: 2
Procedure: Operative attempt at closure — go the operating room to attempt closure
  Arms: 1

SUMMARY:
The hypothesis is that there is no difference between bedside silo placement and operative closure in return of bowel function, ventilator dependence, or length of stay.

The primary outcome variable between the two techniques will be determined from this study that can then be used to develop a definitive study. The likely variables will be length of time to meet discharge criteria, length of hospitalization, time to full feedings, time on mechanical ventilation and total hospital charges.

DETAILED DESCRIPTION:
A strategy of blocked randomization will be utilized. The randomization will be blocked in groups of 4. Randomization sequence will be kept by the principal investigator. After permission is obtained, the next assignment will be obtained. This method assures that the physician obtaining permission will be blind to the treatment group.

The treatment groups will consist of the same medical management, feeding regimen and discharge criteria.

The interventions will be either bedside silo or operative attempt at closure. During attempt at primary closure, the abdomen will be closed completely if the staff anesthesiologist and surgeon agree the belly is not too tight based on ventilatory parameters, vital signs and appearance. If either the surgeon or anesthesiologist should feel the closed abdomen is too tight, a ringed silo will be placed in the operating room, the same silo used in the bedside treatment arm, and the child will continue in the study. When a silo is placed either in the operating room due to inability to close the abdomen or at the bedside, they will be managed the same way. The skin will be dressed in the standard fashion (betadine jelly, xeroform and kerlix). The dressing allows visualization of the bowel. No reductions will be done the day of placement. After one night of observation a tie will be gently placed to apply downward pressure on the bowel. This pressure will not be allowed to increase the peak ventilator pressure by more than 2 cm H2O. One tie will be placed each subsequent day until the tie is within 2 cm of the skin at which point the patient will be scheduled for operative closure the day following the placement of the tie.

The medical management is controlled for resuscitation, sedation, ventilation and feeding between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastroschisis

Exclusion Criteria:

* Born prior to 34 weeks estimated gestational age
* Another congenital anomaly influencing the respiratory status, gastrointestinal status, or the length of hospitalization and recovery.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
this is a pilot study therefore there is no primary outcome variable | 1 year

SECONDARY OUTCOMES:
Time to full feeds, time of ventilation, hospital charges, total time in the operating room, number of operations, fluid resuscitation, total transfusion volume, fluid re | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No